CLINICAL TRIAL: NCT04348721
Title: ASSESSMENT OF COMPLEXITY AND TECHNICAL DIFFICULTIES IN LIVER TRANSPLANTATION: INTERNATIONAL SURVEY OF EXPERTS
Brief Title: INTERNATIONAL SURVEY ON COMPLEXITY IN LIVER TRANSPLANTATION
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Pitié-Salpêtrière Hospital (Other)
Responsible Party: Principal Investigator, Olivier Scatton, Professor, Pitié-Salpêtrière Hospital
Other Study IDs: Pitié-Salpêtrière Hospital
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Liver Transplantation
Keywords: complexity; international survey; surgical difficulty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: online survey — An online survey including 8 case-vignettes was sent to international liver transplant surgeons who had published on liver transplantation. The first part is related to surgeon's own experience. In the second part, the surgeons were asked to rate the difficulty of various situations in liver transplantation on a scale of 1 to 10 (level 1 was labeled as "easier," and level 10 was labeled as "difficult"). In the third part, 8 case-vignettes corresponding to 8 clinical real-life situations are submitted to experts

SUMMARY:
The aim of this study is to perform an online survey to assess the perception of international liver transplant surgeons regarding the complexity and surgical difficulty in liver transplantation and to develop a complexity score and classification.

ELIGIBILITY:
Inclusion Criteria:

* surgeons in liver transplantation center
* all countries

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: International liver transplant surgeons who had published on liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
Identify preoperative criteria to evaluate the degree of technical difficulty during a liver transplantation. | five minuts

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié-Salpêtrière Hospital, APHP, Paris, France

REFERENCES:
- [Background] Lee MK 4th, Gao F, Strasberg SM. Perceived complexity of various liver resections: results of a survey of experts with development of a complexity score and classification. J Am Coll Surg. 2015 Jan;220(1):64-9. doi: 10.1016/j.jamcollsurg.2014.09.017. Epub 2014 Oct 15. PMID 25451665
- [Background] Lee MK 4th, Gao F, Strasberg SM. Completion of a Liver Surgery Complexity Score and Classification Based on an International Survey of Experts. J Am Coll Surg. 2016 Aug;223(2):332-42. doi: 10.1016/j.jamcollsurg.2016.03.039. Epub 2016 Apr 9. PMID 27072308
- [Background] Manceau G, Benoist S, Panis Y, Rault A, Mathonnet M, Goere D, Tuech JJ, Collet D, Penna C, Karoui M. Elective surgery for tumours of the splenic flexure: a French inter-group (AFC, SFCD, FRENCH, GRECCAR) survey. Tech Coloproctol. 2020 Feb;24(2):191-198. doi: 10.1007/s10151-019-02143-2. Epub 2020 Jan 14. PMID 31939046
- [Background] Reames BN, Blair AB, Krell RW, Groot VP, Gemenetzis G, Padussis JC, Thayer SP, Falconi M, Wolfgang CL, Weiss MJ, Are C, He J. Management of Locally Advanced Pancreatic Cancer: Results of an International Survey of Current Practice. Ann Surg. 2021 Jun 1;273(6):1173-1181. doi: 10.1097/SLA.0000000000003568. PMID 31449138